CLINICAL TRIAL: NCT05772416
Title: Diagnostic Value of the Neonatal Neurological Examination to Detect Infants at Risk for Neurological Abnormalities
Brief Title: Neonatal Neurological Examination to Detect Infants at Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4313
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Neonatal Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to establish the diagnostic vcalue of a structured neurological examination to detect eraly neurological abnormlaities in infants at risk of neurological abnormlaiyies.

DETAILED DESCRIPTION:
The study aims to establish the diagnostic vcalue of a structured neurological examination to detect eraly neurological abnormlaities in infants at risk of neurological abnormlaiyies.

Infants at risk of neurological abnormlaiyies, such as very pèretrm infants and infants with asphyxia or with overt neyurologocal abnormla signs suh as convilsions will be assessed with a structured neurological examination and followed over time.

ELIGIBILITY:
Inclusion Criteria:

all newborns with neonatal encephaolopathy or at risk for neurological abnormlaities, such as preterm infants born below 34 weeks or those with convusions

Exclusion Criteria:

families unwilling to sign consent

Ages: 6 Hours to 1 Week | Sex: All
Age Groups: Child
Study Population: all newborns with neonatal encephaolopathy or at risk for neurological abnormlaities, such as preterm infants born below 34 weeks or those with convusions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Hammersmith Neonatal and infant Neurological examination | 5 years
  neurological examination witha score from 0 to 75 with 75 indicating best performance

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, Principal Investigator — F Policlinico Gemelli IRCCS
Locations (1):
- Policlinico gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
only aggregate data as from consensus